CLINICAL TRIAL: NCT03594006
Title: University of Hawai'i Cancer Center Cancer Care Delivery Research: Validation of an Oncology-specific Instrument to Measure Care Coordination
Brief Title: Validation of an Oncology-specific Instrument to Measure Care Coordination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Holcombe-2018-1
Record Dates: First submitted 2018-02-25; First posted 2018-07-20 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Oncology
Keywords: Active Therapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cancer patients on active therapy (Other)
  Interventions: Behavioral: CCI; cancer care coordination instrument

INTERVENTIONS:
Behavioral: CCI; cancer care coordination instrument — Designed to assess cancer patients' perceptions of care coordination

SUMMARY:
The overarching goal of the project is to use a mixed-methods research design to assess the validity of a new instrument developed to assess cancer patients' perceptions of care coordination across varied care settings.

DETAILED DESCRIPTION:
This proposed cancer care delivery research project aims to validate a new instrument (CCI; cancer care coordination instrument) designed to assess cancer patients' perceptions of care coordination. Care coordination (CC) is important for all patients, and it is especially important for cancer patients as they have complex episodes of care, multi-disciplinary interventions, prolonged duration of care, and an overall high symptom burden. Further, CC is critical for cancer patients due to several transition points between stages of care (diagnosis, treatment, survivorship, and end of life), varied settings of care (inpatient, ambulatory), and multiple physicians (medical, surgical, radiation oncologists) and other healthcare providers (e.g., oncology nurses, primary care physicians, physicians/nurses' assistants) providing care.

A CCI validated in ethnically/racially diverse samples can be utilized to identify potential targets for intervention and improvement in CC for specific populations and to reduce or eliminate the disparities in cancer health outcomes. Validation of the CCI under this proposal will have widespread applicability to oncology care across varied practice environments and will form a foundation for the creation of similar tools for other chronic and complex conditions.

ELIGIBILITY:
Inclusion Criteria:

* Active therapy for cancer, defined as a minimum of three exams or therapy visits over a preceding three-month period.
* Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Assessing focus group initial perceptions of the care coordination instrument (CCI) as measured by the participants' Likert scale responses to the instruments' questionnaire items. | 12 months
  We will assess focus group initial perceptions of the care coordination instrument (CCI) as measured by the participants' Likert scale responses to the instruments' questionnaire items. These 27 survey items are used to assess three domains of care coordination. These domains include patient/physician communications, operations and navigation.
  Additionally, the taped narratives and comments of participants provided during the focus group discussions are used to identify and analyze sources of response error in the questionnaire by identifying the cognitive processes respondents use to answer the survey questions. Specifically, whether subjects understand the survey items as intended by the research team.

SECONDARY OUTCOMES:
Assessing patient perceptions of care coordination as measured by the care coordination instrument (CCI). | 12 months
  Secondary outcome measures are cancer patients' perceptions of CC as measured by the CCI. The current proposed CCI contains 27 multiple-choice questions and measures cancer patients' perceptions of four areas of coordination (patient-physician; between health providers; during inpatient-to-ambulatory care transitions; during transitions across different phases of care) that cover three critical domains of CC (Communication, Operational, Navigation).
  Reporting of study results will follow guidelines for qualitative research outlined in the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) Statement and Standard for reporting qualitative research (O'Brien, 2014). The criteria for interviews and focus groups, COREQ, will be followed (Tong et al., 2007). Reported data will include characteristics of the research team and details outlining the theoretical framework, participant selection, setting of the research, and procedures for data collection.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hawaii Cancer Center, Honolulu, Hawaii, United States

REFERENCES:
- [Background] Okado I, Cassel K, Pagano I, Holcombe RF. Development and psychometric evaluation of a questionnaire to measure cancer patients' perception of care coordination. BMC Health Serv Res. 2020 Jan 21;20(1):52. doi: 10.1186/s12913-020-4905-4. PMID 31964391